CLINICAL TRIAL: NCT00418639
Title: Randomized, Double-Blind, Placebo-Controlled Study of Nitazoxanide in the Treatment of Chronic Hepatitis C
Brief Title: Study of Nitazoxanide in the Treatment of Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RM01-3027
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2007-01-05 (Estimated); Status verified 2007-01

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide

SUMMARY:
This study will evaluate the effect of treatment with 24 weeks nitazoxanide monotherapy on end of treatment virologic response, sustained virologic response, reduction of quantitative serum HCV RNA, changes in ALT and safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Chronic hepatitis C infection (at least 6 months) evidenced by a positive enzyme immunoassay for anti-HCV-antibodies and a positive quantitative RT-PCR amplification of HCV RNA.
* Chronic inflammation on liver biopsy compatible with a diagnosis of chronic viral hepatitis.

Exclusion Criteria:

* Patients unable to take oral medications.
* Use of interferon alpha within 90 days or ribavirin within 30 days prior to enrollment.
* Females of child bearing age who are either pregnant, breast-feeding or not using birth control and are sexually active.
* Any investigational drug therapy within 30 days prior to enrollment.
* Patients with other causes of liver disease.
* Patients co-infected with hepatitis A virus, hepatitis B virus or hepatitis D virus based on enzyme immunoassay.
* Patients with history of alcoholism or with an alcohol consumption of >40 grams per day.
* Patients who are clinically unstable.
* Patients with any concomitant condition that, in the opinion of the investigator would preclude evaluation of response or make it unlikely that the contemplated course of therapy and follow-up could be completed.
* History of hypersensitivity or intolerance to nitazoxanide or any of the excipients comprising the nitazoxanide tablets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-02

PRIMARY OUTCOMES:
Virologic response

SECONDARY OUTCOMES:
Sustained virologic response
Quantitative serum HCV RNA
Changes in ALT

CONTACTS AND LOCATIONS:
Overall Officials: Samir M Kabil, MD, Principal Investigator — Cairo Liver & GIT Center; Yehia El-Gohary, MD, Principal Investigator — Department of Tropical Medicine & Infectious Diseases, Alexandria University; Asem Elfert, MD, Principal Investigator — Department of Tropical Medicine & Infectious Diseases, Tanta University School of Medicine
Locations (3):
- Egypt (3):
  - Department of Tropical Medicine & Infectious Diseases, Alexandria University, Alexandria
  - Cairo Liver & GIT Center, Cairo
  - Department of Tropical Medicine & Infectious Diseases, Tanta University School of Medicine, Tanta